CLINICAL TRIAL: NCT06680154
Title: Gamma Oscillations and Working Memory Following Combined 40Hz tACS and iTBS
Brief Title: Induction and Stabilization of Gamma Oscillations With 40 Hz External Brain Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The National Brain Mapping Laboratory (NBML) (Other)
Collaborators: Leibniz Research Centre for Working Environment and Human Factors (Other)
Responsible Party: Principal Investigator, Mohammad Ali Salehinejad, Dr Mohammad Ali Salehinejad, Technical University of Dortmund
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: IfADo_196
Record Dates: First submitted 2024-11-05; First posted 2024-11-08 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Alzheimer Disease; Working Memory; EEG Brain Oscillations
Keywords: Alzheimer's disease; Gamma oscillations; EEG; Transcranial alternating current stimulation, tACS; Intermittent theta burst stimulation
MeSH Terms: conditions — Alzheimer Disease | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Transcranial alternating current stimulation (Active Comparator): During tACS, an alternating electrical current with a 1 milliamp peak-to-peak amplitude will be delivered, featuring a 15-second ramp-up at the start and a 15-second ramp-down at the end. The stimulation duration is 20 minutes and four channels are used for delivering sinusoidal alternating currents to the head. The alternating current was delivered to the prefrontal cortex bilaterally with the electrodes at F3 and F4 and the return electrodes were placed at the ipsilateral mastoids at TP9 and TP10 (international 10-20 EEG electrode placement system).
  Interventions: Device: Transcranial alternating current stimulation
- intermittent theta burst stimulation (Active Comparator): The intermittent theta burst stimulation (iTBS) is regarded as safe for high-frequency neuromodulation. The pulse bursts are applied for two seconds in 5Hz intervals followed by an eight-second break before the next bursts are applied. This pattern is repeated for 190 seconds resulting in 600 pulses per protocol. 80% of the individual subjects' active motor threshold (AMT) are used for stimulation intensity and will be applied four times within a 20-minute time frame starting at 0 minutes, 5 minutes, 10 minutes, and 15 minutes from the beginning of the intervention resulting in 2400 delivered pulses for the whole intervention
  Interventions: Device: Theta burst stimulation
- combited iTBS- tACS peak (Active Comparator): To combine tACS and the iTBS protocol, a customized circuit is developed in-house to phase-lock the TMS pulses to the waveform generated by tACS. TMS pulses were delivered using two figure-of-eight shaped coils (double 70 mm, PMD coil type; Mag and More GmbH, Munich, Germany). For the stimulation, the center of the TMS coils are placed over the two prefrontal tACS electrodes (F3 and F4 electrode positions) with an orientation of 45 degrees to the midline and the handles pointing backward. Using the customized circuit, TMS pulses will be delivered at the peak of the tACS wave.
  Interventions: Device: Transcranial alternating current stimulation; Device: Theta burst stimulation
- Combined iTBS-tACS trough (Active Comparator): To combine tACS and the iTBS protocol, a customized circuit is developed in-house to phase-lock the TMS pulses to the waveform generated by tACS. TMS pulses were delivered using two figure-of-eight shaped coils (double 70 mm, PMD coil type; Mag and More GmbH, Munich, Germany). For the stimulation, the center of the TMS coils are placed over the two prefrontal tACS electrodes (F3 and F4 electrode positions) with an orientation of 45 degrees to the midline and the handles pointing backward. Using the customized circuit, TMS pulses will be delivered at the trough of the tACS wave.
  Interventions: Device: Transcranial alternating current stimulation; Device: Theta burst stimulation
- sham (Sham Comparator): 80% of the individual subjects' active motor threshold (AMT) four times within a 20-minute time frame starting at 0 minutes, 5 minutes, 10 minutes, and 15 minutes from the beginning of the intervention resulting in 2400 delivered pulses for the whole intervention
  Interventions: Device: Sham (No Treatment)

INTERVENTIONS:
Device: Transcranial alternating current stimulation — Transcranial alternating current was delivered utilizing a Starstim 8-channel constant current, battery-powered electric stimulator (Neuroelectrics, Barcelona, Spain). Circular carbon rubber electrodes (2cm radius, 12,57 cm2) were used throughout the stimulation. Before placing the electrodes on the head, the subject's hair was moved to the side
  Arms: Combined iTBS-tACS trough; Transcranial alternating current stimulation; combited iTBS- tACS peak
Device: Theta burst stimulation — the intermittent theta burst stimulation (iTBS) which is regarded as safe for high-frequency neuromodulation. Compared to classical rTMS, where pulses are applied repeatedly at a fixed frequency, iTBS consists of bursts of pulse triplets. In the classical protocol, the bursts are applied for two seconds in 5Hz intervals followed by an eight-second break, before the next bursts are applied. This pattern is repeated for 190 seconds resulting in 600 pulses per protocol.
  Arms: Combined iTBS-tACS trough; combited iTBS- tACS peak; intermittent theta burst stimulation
Device: Sham (No Treatment) — In the case of sham TMS, two different sham coils (double 70mm pCool-SHAM coil, Mag&More GmbH, Munich, Germany) will produce audible clicks at the decibel intensity corresponding to an active coil without the induction of an electromagnetic pulse. Sham tACS will be applied by only ramping the current for 15 seconds up and 15 seconds down at the beginning and end of the stimulation respectively.
  Arms: sham

SUMMARY:
The goal of the present studies is to develop and validate novel stimulation protocols for the entrainment of gamma oscillations, which are associated with many cognitive functions and critically involved in cognitive impairment such as Alzheimer's disease. In this proposal, combination of repetitive transcranial magnetic stimulation (rTMS) and transcranial alternating current stimulation (tACS), which has been shown effective for the induction, and stabilisation of alpha and theta frequencies in our forgoing studies, will be adopted to the gamma frequency range and applied on prefrontal regions as well as model-based cortical areas to enhance and stabilize gamma oscillations, thereby facilitating cognition

DETAILED DESCRIPTION:
Neuropsychiatric disorders are a leading cause of global disability-adjusted life years, and treatment solutions are lacking. Recent findings suggest that non-invasive brain stimulation may be a valuable option in conditions such as epilepsy or Alzheimer's disease (AD). Still, a better understanding of mechanisms and patient-specific factors is needed. Personalized hybrid brain models uniting the physics of electromagnetism with physiology - NeuroTwins (NeTs) - are poised to play a fundamental role in understanding and optimizing the effects of stimulation at the individual level. The purpose of this project is to deliver solutions through model-driven, individualized therapy. A computational framework - weaved and validated across scales and levels of detail - will be proposed to represent the mechanisms of interaction of electric fields with brain networks and assimilate neuroimaging data. This will allow us to characterize the dynamical landscape of the individual brain and define strategies to restore healthy dynamics. The work package, which will take place at IfADo, is part of the consortium collaborating with labs across Europe and USA, aiming to validate and optimize the realistic hybrid brain models developed by NeTs. The targeted subject groups of the IfADo project will be healthy young and old participants. Non-invasive brain stimulation including repetitive transcranial magnetic stimulation and transcranial alternating current stimulation will be applied with electroencephalography, and magnetic resonance spectroscopy as outcome measures. The results are to be translated into a technology pipeline for the design of new personalized neuromodulation protocols which will further be tested in a cohort of AD patients by another clinical consortium member, delivering model-driven breakthroughs in basic and clinical neuroscience, with patients ultimately benefiting from safe, individualized therapy solutions.

ELIGIBILITY:
Inclusion Criteria:

* normal or corrected to normal eye vision
* right-handed
* non-smokers
* being 18-60 years old
* providing written informed consent

Exclusion Criteria:

* history of neurological or psychiatric disorders including seizures or epilepsy,
* Taking CNS medication
* having metal implants
* current pregnancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-07-13 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Working Memory behavioral performance | During procedure (20 minutes)
  Participants view a continuous sequence of alphabet letters, presented as stimuli in Arial font, size 120pt, on a tube screen positioned at 60cm eye distance. The stimuli are shown with a time interval of two seconds between them. The task consisted of six blocks with 70 stimuli, including 12 possible hit trials. Participants were instructed to press the left key on a response box if the presented stimulus matched either the one presented one trial prior (1-Back) or three trials prior (3-Back). In all other cases, participants press the right key. The left button is pressed with the index finger, while the right button is pressed with the middle finger of the right hand, with buttons aligned horizontally. The response condition varied by block, with three blocks for 3-Back and three for 1-Back, and the order was counterbalanced across participants and sessions.
electroencephalogram (EEG) oscillatory power | up to 2 hours after the intervention
  Change in the EEG power in alpha, delta, theta and beta bands
electroencephalogram (EEG) functional connectivity | up to 2 hours after the intervention
  Change in EEG functional connectivity, specifically global efficiency, coherence, and phase-locking value.

CONTACTS AND LOCATIONS:
Locations (1):
- Leibniz-Institut für Arbeitsforschung, Dortmund, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: Undecided